CLINICAL TRIAL: NCT03061890
Title: Developmental Impact of Neonatal Intensive Care Unit (NICU) Exposures: Environmental Influences on Child Health Outcomes (ECHO)
Brief Title: Developmental Impact of NICU Exposures (DINE)
Acronym: DINE
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Judy Aschner, Professor of Pediatrics, Albert Einstein College of Medicine
Other Study IDs: 2016-7369; UG3OD023320 (NIH); UH3OD023320 (NIH)
Record Dates: First submitted 2017-02-03; First posted 2017-02-23 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Prematurity
Keywords: children's environmental health; prematurity; preterm birth; phthalates; NICU; stress; lung health; neurodevelopment; growth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — Urine, hair, teeth, blood, saliva for DNA (optional) samples retained, with potential for extraction of DNA from saliva with separate consent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prematurity and Respiratory Outcomes Program (PROP): extant, NIH-supported preterm birth cohort NCT01435187
- Trial of Late Surfactant (TOLSURF): extant, NIH-supported preterm birth cohort NCT01022580
- NICU Hospital Exposures and Long-Term Health (NICU-HEALTH): extant, NIH-supported preterm birth cohort NCT01963065
- Preterm Erythropoietin Neuroprotection Trial (PENUT): extant, NIH-supported preterm birth cohort NCT01378273

SUMMARY:
The DINE study will test the hypothesis that potentially avoidable NICU-based exposures contribute to the neuro-cognitive and somatic impairments prevalent among NICU graduates. This hypothesis is drawn from the documented impact of phthalate exposure on early development in term-born children, and the acknowledged presence of these toxic chemicals in the NICU. Third trimester in utero exposure to phthalates have been linked to poorer childhood performance in cognition, motor function, attention, hyperactivity and social behavior. Phthalate exposure is also associated with altered onset of puberty and asthma. The multi-site cohort and approach will clarify the role of NICU-based phthalate exposure on high-prevalence clinical outcomes.

DETAILED DESCRIPTION:
Background: Each year in the United States, over 300,000 preterm infants are admitted to neonatal intensive care units (NICUs) where they are exposed to a chemical-intensive hospital environment during a developmentally vulnerable period. Many life-saving and supportive respiratory, nutritional, hematologic and pharmaceutical therapies in the NICU expose preterm infants to potentially harmful chemicals during a life stage analogous to the third trimester of gestation. The NIH-funded DINE study capitalizes on the infrastructure, biorepositories, and extensive clinical databases of four existing preterm cohorts to explore the hypothesis that early life exposure to phthalates adversely impacts neurodevelopment, lung function, growth, adiposity, and pubertal development in childhood.

The scientific premise of the DINE study is that early life exposure to phthalates, a class of chemical plasticizers ubiquitous in the NICU, has long-lasting harmful effects on child health and development, and that these harmful effects are magnified in children born preterm. This premise is based on strong evidence of multisystem adverse health effects in term-born children who are exposed to phthalates in utero during the third trimester of pregnancy or in early infancy. In preterm infants, however, rigorously obtained data on the health effects of phthalates are scant. Dermal, inhalational and intravenous exposures to phthalates are widespread in some NICUs, where preterm infants are cared for during the sensitive "third trimester" developmental window. Moreover, premature infants experience a high prevalence of the adverse health effects that are associated with early life exposures to phthalates in term-born children, including altered neurodevelopment, poor pulmonary function, and maladapted growth. A rigorous, well-designed, sufficiently powered study of NICU-based phthalate exposures and long-term health outcomes of preterm infants has the potential to change care practices, promote regulatory policy changes and lead to mitigation of phthalate exposures in the NICU.

Significance: The proposed research is expected to identify modifiable sources of developmental risk for NICU patients that can inform and improve hospital care and long-term outcome. Moreover, our findings could lead to relatively inexpensive NICU interventions, such as use of non-phthalate containing medical materials, dosing guidelines for elemental metals and guidance for parents and staff on infant stress-reduction, and policy changes (e.g. regulation of the phthalates used in medical devices or changes to the trace metal content of parenteral nutrition) with significant positive potential impacts on life-long morbidities common among NICU graduates. Information gleaned from studying our highly-exposed, highly-vulnerable population may elucidate health impacts of early life exposures that translate to risk reduction in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Children who were study participants in one of the four extant preterm cohorts (PROP, TOLSURF, NICU-HEALTH, and PENUT) that comprise the combined DINE cohort and who were followed to study endpoint at one of the clinical sites in DINE.
* Newly recruited preterm infants admitted to the NICU at the Icahn School of Medicine at Mount Sinai
* Newly recruited preterm and term infants who participated in the PRISM study at University of Rochester
* Parents agreed to be re-contacted or local Institutional Review Board (IRB) grants permission to recontact families to obtain consent to participate in DINE.

Exclusion Criteria:

* Family requested that they not be contacted after their child completed the parent study
* Family is unlikely to be available for long-term follow-up

Max Age: 12 Years | Sex: All
Age Groups: Child
Study Population: Former preterm infants who were participants hospitalized in the NICU of one of the 8 clinical sites participating in the UH3 phase of the ECHO and DINE studies and whose parents had consented to participate in one of the 4 extent cohorts of the following NIH-supported studies: Prematurity and Respiratory Outcomes Program (PROP), the Trial of Late Surfactant (TOLSURF), the NICU Hospital Exposures and Long-Term Health (NICU-HEALTH) study and the Preterm Erythropoietin Neuroprotection Trial (PENUT) study and agreed to longitudinal follow up of infants as part of DINE
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Association between NICU environmental exposures and lung health and asthma measured by Brief Respiratory Questionnaire | One time between the ages of 3 to 4
  Brief Respiratory Questionnaire to determine association between exposure and lung health
Associations between NICU environmental exposures and lung health and asthma measured by the PROMIS® (Patient-Reported Outcomes Measurement Information System) Parent Proxy Asthma Impact item bank | One time between the ages of 5 to 6
  PROMIS® (Patient-Reported Outcomes Measurement Information System) Parent Proxy Asthma Impact item bank to determine association between exposure and asthma
Associations between NICU environmental exposures and lung health and asthma measured by PhenX (consensus measures for Phenotypes and eXposures) Toolkit measures of spirometry and bronchodilator responsiveness | Twice between the ages of 8 to 12
  PhenX (consensus measures for Phenotypes and eXposures) Toolkit measures of spirometry and bronchodilator responsiveness to determine association between exposure and asthma
Associations between NICU environmental exposures and lung health and asthma measured by the PROMIS Pediatric Asthma Impact item bank. | Twice between the ages of 8 to 12
  PROMIS Pediatric Asthma Impact item bank to determine the association between exposures and asthma
Associations between NICU environmental exposures and neurocognitive behavioral development measured by NIH Toolbox Early Childhood Cognition Battery | Twice within 24 months between the ages of 3 to 5
  NIH Toolbox Early Childhood Cognition Battery to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and neurocognitive behavioral development measured by NIH Toolbox Cognition Battery | Twice within 24 months between the ages of 7 to 9
  NIH Toolbox Cognition Battery to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and neurocognitive behavioral development measured by NIH Toolbox Early Childhood Motor Battery | Twice within 24 months between the ages of 4 to 6
  NIH Toolbox Early Childhood Motor Battery to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and neurocognitive behavioral development measured by NIH Toolbox Motor Battery | Twice between the ages of 8 to 12
  NIH Toolbox Motor Battery to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and neurocognitive behavioral development measured by Child Behavior Checklist (CBCL) | One time between the ages of 3 to 4
  Child Behavior Checklist (CBCL) to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and neurocognitive behavioral development measured by PROMIS Cognitive Item bank | Three times between the ages of 5 to 12
  PROMIS Cognitive Item bank to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and neurocognitive behavioral development measured by PROMIS Pediatric Mobility Item bank | Three times between the ages of 5 to 12
  PROMIS Pediatric Mobility Item bank to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and neurocognitive behavioral development measured by PROMIS Pediatric Upper Extremity Item bank | Three times between the ages of 5 to 12
  PROMIS Pediatric Upper Extremity Item to determine the associations between exposures and neurocognitive behavioral development
Associations between NICU environmental exposures and growth and obesity as measured by height, weight, head circumference, mid-upper arm circumference and bioimpedence | Annually, up to 12 years
  Measurement of height, weight, head circumference, mid-upper arm circumference and bioimpedence scale to determine associations between exposures and heathy growth and obesity
Associations between NICU environmental exposures and growth and obesity as measured by parent report height and weight | Annually, up to 12 years
  Parent reported height and weight to determine associations between exposures and healthy growth and obesity
Associations between NICU environmental exposures and pubertal development measured by PhenX Assessment of Pubertal Development | Annually, up to 12 years
  PhenX Assessment of Pubertal Development to determine associations between exposures and pubertal development

CONTACTS AND LOCATIONS:
Overall Officials: Judy L Aschner, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (11):
- United States (11):
  - University of Florida, Jacksonville, Florida
  - National Institute for Children's Health Quality, Boston, Massachusetts
  - Children's Health Care, Inc., Minneapolis, Minnesota
  - University at Buffalo State University of New York, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester, Rochester, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
All efforts, within reason, are made to keep protected health information (PHI) private, including data gathered for research studies. Using or sharing ("disclosure") such data must follow federal privacy rules. All PHI about children in the study will be entered into REDCap, a secure, web-based data collection platform. Study patients will be identified only by a study identification (ID) number. Access to the REDCap study database is restricted to study personnel, password protected and behind a Medical Center firewall. The study child's name and medical record number will appear only on the Screening Log which contains no other PHI. Only the study team will have access to the Screening Log.

REFERENCES:
- [Background] Aschner JL, Bancalari EH, McEvoy CT. Can We Prevent Bronchopulmonary Dysplasia? J Pediatr. 2017 Oct;189:26-30. doi: 10.1016/j.jpeds.2017.08.005. No abstract available. PMID 28947055
- [Background] Wright RO, Teitelbaum S, Thompson C, Balshaw D; CHEAR Network. The child health exposure analysis resource as a vehicle to measure environment in the environmental influences on child health outcomes program. Curr Opin Pediatr. 2018 Apr;30(2):285-291. doi: 10.1097/MOP.0000000000000601. PMID 29406438
- [Background] Zhang X, Smith N, Spear E, Stroustrup A. Neighborhood characteristics associated with COVID-19 burden-the modifying effect of age. J Expo Sci Environ Epidemiol. 2021 May;31(3):525-537. doi: 10.1038/s41370-021-00329-1. Epub 2021 May 4. PMID 33947953
- [Result] Stroustrup A, Teitelbaum SL, Aschner JL. The Value of Preterm Infant Environmental Health Cohorts: The Canary in the Coal Mine. JAMA Pediatr. 2017 Dec 1;171(12):1139-1140. doi: 10.1001/jamapediatrics.2017.3230. No abstract available. PMID 29059271
- [Result] Stroustrup A, Bragg JB, Andra SS, Curtin PC, Spear EA, Sison DB, Just AC, Arora M, Gennings C. Neonatal intensive care unit phthalate exposure and preterm infant neurobehavioral performance. PLoS One. 2018 Mar 5;13(3):e0193835. doi: 10.1371/journal.pone.0193835. eCollection 2018. PMID 29505594
- [Result] Stroustrup A, Bragg JB, Busgang SA, Andra SS, Curtin P, Spear EA, Just AC, Arora M, Gennings C. Sources of clinically significant neonatal intensive care unit phthalate exposure. J Expo Sci Environ Epidemiol. 2020 Jan;30(1):137-148. doi: 10.1038/s41370-018-0069-2. Epub 2018 Sep 21. PMID 30242269
- [Result] Conradt E, Flannery T, Aschner JL, Annett RD, Croen LA, Duarte CS, Friedman AM, Guille C, Hedderson MM, Hofheimer JA, Jones MR, Ladd-Acosta C, McGrath M, Moreland A, Neiderhiser JM, Nguyen RHN, Posner J, Ross JL, Savitz DA, Ondersma SJ, Lester BM. Prenatal Opioid Exposure: Neurodevelopmental Consequences and Future Research Priorities. Pediatrics. 2019 Sep;144(3):e20190128. doi: 10.1542/peds.2019-0128. PMID 31462446
- [Result] Tylavsky FA, Ferrara A, Catellier DJ, Oken E, Li X, Law A, Dabelea D, Rundle A, Gilbert-Diamond D, Hivert MF, Breton CV, Cassidy-Bushrow AE, Mueller NT, Hunt KJ, Arteaga SS, Lombo T, Mahabir S, Ruden D, Sauder K, Hedderson MM, Zhu Y, Polk S, Mihalopoulos NL, Vos M, Pyles L, Roary M, Aschner J, Karagas MR, Trasande L. Understanding childhood obesity in the US: the NIH environmental influences on child health outcomes (ECHO) program. Int J Obes (Lond). 2020 Mar;44(3):617-627. doi: 10.1038/s41366-019-0470-5. Epub 2019 Oct 24. PMID 31649277
- [Result] Pourkaviani S, Zhang X, Spear EA, D'Agostino M, Satty RE, Liu SH, Stroustrup A. Clinical validation of the Neonatal Infant Stressor Scale with preterm infant salivary cortisol. Pediatr Res. 2020 Jun;87(7):1237-1243. doi: 10.1038/s41390-019-0713-0. Epub 2019 Dec 17. PMID 31847006
- [Result] Stroustrup A, Bragg JB, Spear EA, Aguiar A, Zimmerman E, Isler JR, Busgang SA, Curtin PC, Gennings C, Andra SS, Arora M. Cohort profile: the Neonatal Intensive Care Unit Hospital Exposures and Long-Term Health (NICU-HEALTH) cohort, a prospective preterm birth cohort in New York City. BMJ Open. 2019 Nov 25;9(11):e032758. doi: 10.1136/bmjopen-2019-032758. PMID 31772104
- [Result] Faro EZ, Sauder KA, Anderson AL, Dunlop AL, Kerver JM, McGrath M, Roary M, Roman CW, Weidinger C, Huddleston KC. Characteristics of Environmental influences on Child Health Outcomes (ECHO) Cohorts Recruited During Pregnancy. MCN Am J Matern Child Nurs. 2021 Jul-Aug 01;46(4):230-235. doi: 10.1097/NMC.0000000000000725. PMID 33993167
- [Result] Schantz SL, Eskenazi B, Buckley JP, Braun JM, Sprowles JN, Bennett DH, Cordero J, Frazier JA, Lewis J, Hertz-Picciotto I, Lyall K, Nozadi SS, Sagiv S, Stroustrup A, Volk HE, Watkins DJ; program collaborators for Environmental influences on Child Health Outcomes. A framework for assessing the impact of chemical exposures on neurodevelopment in ECHO: Opportunities and challenges. Environ Res. 2020 Sep;188:109709. doi: 10.1016/j.envres.2020.109709. Epub 2020 May 23. PMID 32526495
- [Result] Zhang X, Spear E, Gennings C, Curtin PC, Just AC, Bragg JB, Stroustrup A. The association of prenatal exposure to intensive traffic with early preterm infant neurobehavioral development as reflected by the NICU Network Neurobehavioral Scale (NNNS). Environ Res. 2020 Apr;183:109204. doi: 10.1016/j.envres.2020.109204. Epub 2020 Jan 31. PMID 32311904
- [Result] Stratakis N, Garcia E, Chandran A, Hsu T, Alshawabkeh A, Aris IM, Aschner JL, Breton C, Burbank A, Camargo CA Jr, Carroll KN, Chen Z, Claud EC, Dabelea D, Dunlop AL, Elliott AJ, Ferrara A, Ganiban JM, Gern JE, Gold DR, Gower WA, Hertz-Picciotto I, Karagas MR, Karr CJ, Lester B, Leve LD, Litonjua AA, Ludena Y, McEvoy CT, Miller RL, Mueller NT, O'Connor TG, Oken E, O'Shea TM, Perera F, Stanford JB, Rivera-Spoljaric K, Rundle A, Trasande L, Wright RJ, Zhang Y, Zhu Y, Berhane K, Gilliland F, Chatzi L; on behalf of program collaborators for Environmental Influences on Child Health Outcomes. The Role of Childhood Asthma in Obesity Development: A Nationwide US Multicohort Study. Epidemiology. 2022 Jan 1;33(1):131-140. doi: 10.1097/EDE.0000000000001421. PMID 34561347
- [Result] Lyall K, Ning X, Aschner JL, Avalos LA, Bennett DH, Bilder DA, Bush NR, Carroll KN, Chu SH, Croen LA, Dabelea D, Daniels JL, Duarte C, Elliott AJ, Fallin MD, Ferrara A, Hertz-Picciotto I, Hipwell AE, Jensen ET, Johnson SL, Joseph RM, Karagas M, Kelly RS, Lester BM, Margolis A, McEvoy CT, Messinger D, Neiderhiser JM, O'Connor TG, Oken E, Sathyanarayana S, Schmidt RJ, Sheinkopf SJ, Talge NM, Turi KN, Wright RJ, Zhao Q, Newschaffer C, Volk HE, Ladd-Acosta C, Environmental Influences On Child Health Outcomes OBOPCF. Cardiometabolic Pregnancy Complications in Association With Autism-Related Traits as Measured by the Social Responsiveness Scale in ECHO. Am J Epidemiol. 2022 Jul 23;191(8):1407-1419. doi: 10.1093/aje/kwac061. PMID 35362025
- [Result] Knapp EA, Dong Y, Dunlop AL, Aschner JL, Stanford JB, Hartert T, Teitelbaum SL, Hudak ML, Carroll K, O'Connor TG, McEvoy CT, O'Shea TM, Carnell S, Karagas MR, Herbstman JB, Dabelea D, Ganiban JM, Ferrara A, Hedderson M, Bekelman TA, Rundle AG, Alshawabkeh A, Gilbert-Diamond D, Fry RC, Chen Z, Gilliland FD, Wright RJ, Camargo CA, Jacobson L, Lester BM, Hockett CW, Hodges ML, Chandran A; Environmental Influences on Child Health Outcomes. Changes in BMI During the COVID-19 Pandemic. Pediatrics. 2022 Sep 1;150(3):e2022056552. doi: 10.1542/peds.2022-056552. PMID 35768891
- [Result] Roubinov D, Musci RJ, Hipwell AE, Wu G, Santos H, Felder JN, Faleschini S, Conradt E, McEvoy CT, Lester BM, Buss C, Elliott AJ, Cordero JF, Stroustrup A, Bush NR. Trajectories of depressive symptoms among mothers of preterm and full-term infants in a national sample. Arch Womens Ment Health. 2022 Aug;25(4):807-817. doi: 10.1007/s00737-022-01245-5. Epub 2022 Jun 16. PMID 35708790
- [Result] Knapp EA, Kress AM, Parker CB, Page GP, McArthur K, Gachigi KK, Alshawabkeh AN, Aschner JL, Bastain TM, Breton CV, Bendixsen CG, Brennan PA, Bush NR, Buss C, Camargo CA Jr, Catellier D, Cordero JF, Croen L, Dabelea D, Deoni S, D'Sa V, Duarte CS, Dunlop AL, Elliott AJ, Farzan SF, Ferrara A, Ganiban JM, Gern JE, Giardino AP, Towe-Goodman NR, Gold DR, Habre R, Hamra GB, Hartert T, Herbstman JB, Hertz-Picciotto I, Hipwell AE, Karagas MR, Karr CJ, Keenan K, Kerver JM, Koinis-Mitchell D, Lau B, Lester BM, Leve LD, Leventhal B, LeWinn KZ, Lewis J, Litonjua AA, Lyall K, Madan JC, McEvoy CT, McGrath M, Meeker JD, Miller RL, Morello-Frosch R, Neiderhiser JM, O'Connor TG, Oken E, O'Shea M, Paneth N, Porucznik CA, Sathyanarayana S, Schantz SL, Spindel ER, Stanford JB, Stroustrup A, Teitelbaum SL, Trasande L, Volk H, Wadhwa PD, Weiss ST, Woodruff TJ, Wright RJ, Zhao Q, Jacobson LP, Influences On Child Health Outcomes OBOPCFE. The Environmental Influences on Child Health Outcomes (ECHO)-Wide Cohort. Am J Epidemiol. 2023 Aug 4;192(8):1249-1263. doi: 10.1093/aje/kwad071. PMID 36963379
- [Result] Bekelman TA, Knapp EA, Dong Y, Dabelea D, Bastain TM, Breton CV, Carroll KN, Camargo CA, Davis AM, Dunlop AL, Elliott AJ, Ferrara A, Fry RC, Ganiban JM, Gilbert-Diamond D, Gilliland FD, Hedderson MM, Hipwell AE, Hockett CW, Huddleston KC, Karagas MR, Kelly N, Lai JS, Lester BM, Lucchini M, Melough MM, Mihalopoulos NL, O'Shea TM, Rundle AG, Stanford JB, VanBronkhorst S, Wright RJ, Zhao Q, Sauder KA; program collaborators for Environmental influences on Child Health Outcomes (ECHO). Sociodemographic Variation in Children's Health Behaviors During the COVID-19 Pandemic. Child Obes. 2023 Jun;19(4):226-238. doi: 10.1089/chi.2022.0085. Epub 2022 Jul 19. PMID 35856858
- [Result] O'Shea TM, McGrath M, Aschner JL, Lester B, Santos HP Jr, Marsit C, Stroustrup A, Emmanuel C, Hudak M, McGowan E, Patel S, Fry RC; program collaborators for Environmental influences on Child Health Outcomes. Environmental influences on child health outcomes: cohorts of individuals born very preterm. Pediatr Res. 2023 Apr;93(5):1161-1176. doi: 10.1038/s41390-022-02230-5. Epub 2022 Aug 10. PMID 35948605
- [Result] Lucchini M, Bekelman TA, Li M, Knapp EA, Dong Y, Ballard S, Deoni S, Dunlop AL, Elliott AJ, Ferrara A, Friedman C, Galarce M, Gilbert-Diamond D, Glueck D, Hedderson M, Hockett CW, Karagas MR, LeBourgeois MK, Margolis A, McDonald J, Ngai P, Pellerite M, Sauder K, Ma T, Dabelea D; Environmental influences on Child Health Outcomes. Impact of the COVID-19 pandemic on children's sleep habits: an ECHO study. Pediatr Res. 2023 Feb;93(3):586-594. doi: 10.1038/s41390-022-02309-z. Epub 2022 Oct 4. PMID 36195633
- [Result] Aris IM, Perng W, Dabelea D, Padula AM, Alshawabkeh A, Velez-Vega CM, Aschner JL, Camargo CA Jr, Sussman TJ, Dunlop AL, Elliott AJ, Ferrara A, Zhu Y, Joseph CLM, Singh AM, Hartert T, Cacho F, Karagas MR, North-Reid T, Lester BM, Kelly NR, Ganiban JM, Chu SH, O'Connor TG, Fry RC, Norman G, Trasande L, Restrepo B, James P, Oken E; Program Collaborators for Environmental Influences on Child Health Outcomes. Associations of Neighborhood Opportunity and Social Vulnerability With Trajectories of Childhood Body Mass Index and Obesity Among US Children. JAMA Netw Open. 2022 Dec 1;5(12):e2247957. doi: 10.1001/jamanetworkopen.2022.47957. PMID 36547983
- [Result] Nanishi M, Chandran A, Li X, Stanford JB, Alshawabkeh AN, Aschner JL, Dabelea D, Dunlop AL, Elliott AJ, Gern JE, Hartert T, Herbstman J, Hershey GKK, Hipwell AE, Karagas MR, Karr CJ, Leve LD, Litonjua AA, McEvoy CT, Miller RL, Oken E, O'Shea TM, Paneth N, Weiss ST, Wright RO, Wright RJ, Carroll KN, Zhang X, Zhao Q, Zoratti E, Camargo CA Jr, Hasegawa K; Environmental Influences on Child Health Outcomes (ECHO) Investigators. Association of Severe Bronchiolitis during Infancy with Childhood Asthma Development: An Analysis of the ECHO Consortium. Biomedicines. 2022 Dec 22;11(1):23. doi: 10.3390/biomedicines11010023. PMID 36672531
- [Result] Camerota M, McGowan EC, Aschner J, Stroustrup A, Karagas MR, Conradt E, Crowell SE, Brennan PA, Carter BS, Check J, Dansereau LM, DellaGrotta SA, Everson TM, Helderman JB, Hofheimer JA, Kuiper JR, Loncar CM, Marsit CJ, Neal CR, O'Shea TM, Pastyrnak SL, Sheinkopf SJ, Smith LM, Zhang X, Lester BM. Prenatal and perinatal factors associated with neonatal neurobehavioral profiles in the ECHO Program. Pediatr Res. 2023 Aug;94(2):762-770. doi: 10.1038/s41390-023-02540-2. Epub 2023 Feb 25. PMID 36841884
- [Result] Hedderson MM, Bekelman TA, Li M, Knapp EA, Palmore M, Dong Y, Elliott AJ, Friedman C, Galarce M, Gilbert-Diamond D, Glueck D, Hockett CW, Lucchini M, McDonald J, Sauder K, Zhu Y, Karagas MR, Dabelea D, Ferrara A; Environmental Influences on Child Health Outcomes Program. Trends in Screen Time Use Among Children During the COVID-19 Pandemic, July 2019 Through August 2021. JAMA Netw Open. 2023 Feb 1;6(2):e2256157. doi: 10.1001/jamanetworkopen.2022.56157. PMID 36790805
- [Result] Chandran A, Burjak M, Petimar J, Hamra G, Melough MM, Dunlop AL, Snyder BM, Litonjua AA, Hartert T, Gern J, Alshawabkeh AN, Aschner J, Camargo CA Jr, Dabelea D, Duarte CS, Ferrara A, Ganiban JM, Gilliland F, Gold DR, Hedderson M, Herbstman JB, Hockett C, Karagas MR, Kerver JM, Lee-Sarwar KA, Lester B, McEvoy CT, Niu Z, Stanford JB, Wright R, Zimmerman E, Farzan S, Zhang Z, Knapp E. Changes in Body Mass Index Among School-Aged Youths Following Implementation of the Healthy, Hunger-Free Kids Act of 2010. JAMA Pediatr. 2023 Apr 1;177(4):401-409. doi: 10.1001/jamapediatrics.2022.5828. PMID 36780186
- [Result] Moog NK, Cummings PD, Jackson KL, Aschner JL, Barrett ES, Bastain TM, Blackwell CK, Bosquet Enlow M, Breton CV, Bush NR, Deoni SCL, Duarte CS, Ferrara A, Grant TL, Hipwell AE, Jones K, Leve LD, Lovinsky-Desir S, Miller RK, Monk C, Oken E, Posner J, Schmidt RJ, Wright RJ, Entringer S, Simhan HN, Wadhwa PD, O'Connor TG, Musci RJ, Buss C; ECHO collaborators. Intergenerational transmission of the effects of maternal exposure to childhood maltreatment in the USA: a retrospective cohort study. Lancet Public Health. 2023 Mar;8(3):e226-e237. doi: 10.1016/S2468-2667(23)00025-7. PMID 36841563
- [Result] Hofheimer JA, McGrath M, Musci R, Wu G, Polk S, Blackwell CK, Stroustrup A, Annett RD, Aschner J, Carter BS, Check J, Conradt E, Croen LA, Dunlop AL, Elliott AJ, Law A, Leve LD, Neiderhiser JM, O'Shea TM, Salisbury AL, Sathyanarayana S, Singh R, Smith LM, Aguiar A, Angal J, Carliner H, McEvoy C, Ondersma SJ, Lester B; Program Collaborators for Environmental influences on Child Health Outcomes. Assessment of Psychosocial and Neonatal Risk Factors for Trajectories of Behavioral Dysregulation Among Young Children From 18 to 72 Months of Age. JAMA Netw Open. 2023 Apr 3;6(4):e2310059. doi: 10.1001/jamanetworkopen.2023.10059. PMID 37099294
- [Result] Miller RL, Schuh H, Chandran A, Aris IM, Bendixsen C, Blossom J, Breton C, Camargo CA Jr, Canino G, Carroll KN, Commodore S, Cordero JF, Dabelea DM, Ferrara A, Fry RC, Ganiban JM, Gern JE, Gilliland FD, Gold DR, Habre R, Hare ME, Harte RN, Hartert T, Hasegawa K, Khurana Hershey GK, Jackson DJ, Joseph C, Kerver JM, Kim H, Litonjua AA, Marsit CJ, McEvoy C, Mendonca EA, Moore PE, Nkoy FL, O'Connor TG, Oken E, Ownby D, Perzanowski M, Rivera-Spoljaric K, Ryan PH, Singh AM, Stanford JB, Wright RJ, Wright RO, Zanobetti A, Zoratti E, Johnson CC; of program collaborators for Environmental influences on Child Health Outcomes. Incidence rates of childhood asthma with recurrent exacerbations in the US Environmental influences on Child Health Outcomes (ECHO) program. J Allergy Clin Immunol. 2023 Jul;152(1):84-93. doi: 10.1016/j.jaci.2023.03.016. Epub 2023 Mar 25. PMID 36972767
- [Result] McGowan EC, McGrath M, Law A, O'Shea TM, Aschner JL, Blackwell CK, Fry RC, Ganiban JM, Higgins R, Margolis A, Sathyanarayana S, Taylor G, Alshawabkeh AN, Cordero JF, Spillane NT, Hudak ML, Camargo CA Jr, Dabelea D, Dunlop AL, Elliott AJ, Ferrara AM, Talavera-Barber M, Singh AM, Karagas MR, Karr C, O'Connor TG, Paneth N, Wright RJ, Wright RO, Cowell W, Stanford JB, Bendixsen C, Lester BM; program collaborators for Environmental Influences on Child Health Outcomes (ECHO). Health Care Utilization During the COVID-19 Pandemic Among Individuals Born Preterm. JAMA Netw Open. 2023 Apr 3;6(4):e2310696. doi: 10.1001/jamanetworkopen.2023.10696. PMID 37115545
- [Result] Wood CT, Churchill ML, McGrath M, Aschner J, Brunwasser SM, Geiger S, Gogcu S, Hartert TV, Hipwell AE, Lee-Sarwar K, Lyall K, Moog NK, O'Connor TG, O'Shea TM, Smith PB, Wright RJ, Zhang X, Zimmerman E, Huddleston KC, Brown CL; program collaborators for Environmental influences on Child Health Outcomes. Maternal stress and early childhood BMI among US children from the Environmental influences on Child Health Outcomes (ECHO) program. Pediatr Res. 2023 Dec;94(6):2085-2091. doi: 10.1038/s41390-023-02750-8. Epub 2023 Jul 21. PMID 37479746
- [Result] Martenies SE, Zhang M, Corrigan AE, Kvit A, Shields T, Wheaton W, Around Him D, Aschner J, Talavera-Barber MM, Barrett ES, Bastain TM, Bendixsen C, Breton CV, Bush NR, Cacho F, Camargo CA Jr, Carroll KN, Carter BS, Cassidy-Bushrow AE, Cowell W, Croen LA, Dabelea D, Duarte CS, Dunlop AL, Everson TM, Habre R, Hartert TV, Helderman JB, Hipwell AE, Karagas MR, Lester BM, LeWinn KZ, Magzamen S, Morello-Frosch R, O'Connor TG, Padula AM, Petriello M, Sathyanarayana S, Stanford JB, Woodruff TJ, Wright RJ, Kress AM; Program Collaborators for Environmental Influences on Child Health Outcomes. Developing a National-Scale Exposure Index for Combined Environmental Hazards and Social Stressors and Applications to the Environmental Influences on Child Health Outcomes (ECHO) Cohort. Int J Environ Res Public Health. 2023 Jul 10;20(14):6339. doi: 10.3390/ijerph20146339. PMID 37510572
- [Result] Stroustrup A, Zhang X, Spear E, Bandyopadhyay S, Narasimhan S, Meher AK, Choi J, Qi G, Poindexter BB, Teitelbaum SL, Andra SS, Gennings C, Aschner JL. Phthalate exposure in the neonatal intensive care unit is associated with development of bronchopulmonary dysplasia. Environ Int. 2023 Aug;178:108117. doi: 10.1016/j.envint.2023.108117. Epub 2023 Jul 26. PMID 37517179
- See also: NIH Environmental influences on Child Health Outcomes (ECHO) Program — http://www.nih.gov/echo